CLINICAL TRIAL: NCT04628858
Title: Continuous Monitoring of Physiological Parameters for Early Detection of Complications in Postoperative Vascular Surgical Patients - An Observational Study
Brief Title: Wireless Assessment of Respiratory and Circulatory Distress in Vascular Surgical Patients - An Observational Study
Acronym: WARD-VASC
Status: Completed | Type: Observational
Sponsor: Eske Kvanner Aasvang (Other)
Responsible Party: Sponsor-Investigator, Eske Kvanner Aasvang, Dr. Med., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-19086583
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Complication of Surgical Procedure; Complication of Anesthesia; Respiratory Complication; Circulatory; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Troponin-T
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Primary group

SUMMARY:
Vascular postsurgical patients have a high risk of morbidity and mortality. On top of that, patients undergoing vascular surgery usually have a high burden of comorbidities.

After a short stay in the post-operative ward, patients are usually transferred to a standard surgical ward.

Monitoring of physiological parameters by intermittent manual recordings 8-12 hours apart, is today's standard of care in hospitals. However, no effect on length of hospital stay, morbidity or mortality has been proven. This may be due to the up to 12 hours of unobserved time that can occur, where physiological deviations can progress resulting in clinical adverse outcomes such as myocardial infarction or stroke.

Vital sign micro events are occurrences when patient physiological parameters deviates significantly from what can be understood as normal physiology. Since adverse outcomes in patients rarely happens without deviating physiological parameters, it is to be investigated if micro events can be used to predict clinical adverse outcomes to patients. We acknowledge that during the observation period, the number of false alarms should be kept to a minimum to avoid the risk of 'alarm fatigue'

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Copenhagen University Hospital
* Patients with Peripheral Arteriel Disease(PAD)
* Patients undergoing open infraligamentary revascularization
* Emergency or subacute surgery
* Admission the day before surgery, and expected length of stay more than 2 days.

Exclusion Criteria:

* Patient expected not to cooperate
* Patients with dementia or not able to give informed consent
* Patient allergic to plaster, plastic or silicone
* Patients with pacemaker or implantable cardioverter-defibrillator (ICD) unit
* Patients in isolation
* Active therapy withdrawn
* Patients previously included in the other study branches
* Patients with >20 mmHg in difference in systolic blood pressure between the two arms.
* Expected discharge within less than 24 hours from possible inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 patients admitted for elective or subacute vascular surgical intervention, as noted in the inclusion criteria, will be included on the day before their surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Physiologic abnormal vital signs - Cumulative duration | From inclusion until 4 days or discharge
  Cumulative duration of physiologic vital signs within certain thresholds outside normalcy

SECONDARY OUTCOMES:
Physiologic abnormal vital signs - Episodes of sustained duration | From inclusion until 4 days or discharge
  Episodes of sustained duration of physiologic vital signs within certain thresholds outside normalcy, with different minimum durations

OTHER OUTCOMES:
Any serious adverse events | 30 days
  In accordance with ICH-GCP: any untoward medical occurrence that(...)
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Requires intervention to prevent permanent impairment or damage
Readmission | 6 months
ICU admission | 6 months
Mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eske K Aasvang, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No